CLINICAL TRIAL: NCT07073651
Title: Response of Lipid Profile to Virtual Reality Games Versus Moderate Aerobic Exercise Training in Children With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mina Atef Georgui Elias, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014233-8
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Obese Children and Adolescents; Adolescent Obesity; Obesity; Body Mass Index
Keywords: Obesity; Body mass index; Virtual Reality games; aerobic exercise; adolescent obesity; obese children; Moderate intensity aerobic exercise; dietary advices
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exercise (Experimental): The experimental group included 60 adolescent obese children of both genders (class I obesity, BMI: 30-34.99) who received diet advices and virtual reality exercises 5 times per week for 12 weeks. Each participating child started the session with 5 minutes warming up exercises then followed by the main part which was consisted of 30 min of exercise where the child played the game using virtual reality X-Box and did different physical activities that included both the upper and lower extremities according to the game's requirements, and after that a 5 min cool-down part that involved some static flexibility exercise to allow the heart rate to lower, the total session that would be applied about 40 min (including 30 mins of Virtual reality exercises)
  Interventions: Other: Dietary Advices; Other: Virtual reality games exercise
- Moderate intensity aerobic exercise (Active Comparator): This group serves as the control group, it included 60 adolescent obese children of both genders (class I obesity, BMI: 30-34.99) who received diet advice and moderate intensity aerobic exercises (using treadmill training) 5 times per week for 12 weeks. Each participating child started the session with 5 minutes of warming-up exercises. Then the main exercise phase is performed at 50-60% of age-predicted peak heart rate using a treadmill for 30 minutes. Finally, a 5 min cool-down period is allowed, the total session took 40 minutes.
  Interventions: Other: Moderate Intensity Aerobic Exercise; Other: Dietary Advices

INTERVENTIONS:
Other: Moderate Intensity Aerobic Exercise — moderate intensity aerobic exercises (using treadmill training) 5 times per week for 12 weeks. Each participating child started the session with 5 minutes of warming-up exercises. Then the main exercise phase is performed at 50-60% of age-predicted peak heart rate using a treadmill for 30 minutes. Finally, a 5 min cool-down period is allowed, the total session took 40 minutes.
  Arms: Moderate intensity aerobic exercise
Other: Dietary Advices — The Obese adolescent children participated in the study received diet advices based on a balanced low calorie diet (1500 Kcal)
Other: Virtual reality games exercise — Virtual reality games exercises 5 times per week for 12 weeks. Each participating child started the session with 5 minutes warming up exercises then followed by the main part which was consisted of 30 min of exercise where the child played the game using virtual reality X-Box and did different physical activities that included both the upper and lower extremities according to the game's requirements, and after that a 5 min cool-down part that involved some static flexibility exercises to allow the heart rate to lower, the total session that would be applied about 40 min (including 30 mins of Virtual reality exercises)
  Arms: Virtual Reality Exercise

SUMMARY:
This trial is aiming to study the effect of virtual reality video gaming in comparison with moderate intensity aerobic exercises on lipid profile in children with Obesity

DETAILED DESCRIPTION:
The study will assess whether virtual reality games, dietary advices and moderate intensity aerobic exercise lead to significant differences in lipid profile in class I obese adolescent children. Additionally, the study will examine whether these interventions has impacts on the children body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescent children
* age from 11 to 18 years old only.
* Class I Obesity (Body Mass Index from 30 to 34.99 kg/m2)
* Clinically and medically stable
* Without any impairment of sensation or other neurological or psychological problems.

Exclusion Criteria:

* Adolescents with visual and/or auditory defects
* Normal weight adolescent children (Body Mass Index from 18 to 24.99 kg/m2) or below average weight (BMI less than 18 kg/m2) or Class II and III Obesity (BMI above 35 kg/m2)
* Children with significant tightness and/or deformity of upper or lower limbs
* Participants with neurological disorders that affect balance or mentality (e.g. epilepsy).
* Adolescents with advanced radiographic changes include: Bone destruction, Bony ankylosis, Knee joint subluxation, and Epiphysial fracture)
* Any lower limb deformities in the lower limbs.
* Participants with cardiopulmonary diseases.
* Diabetic children or those under insulin therapy, uncontrolled bronchial asthma, anemia, and Pathological causes of obesity (endocrinal, genetic syndromes...etc.).

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Body mass index | From enrollment to the end of treatment at 12 weeks
  It is the weight (in kilograms) divided by the height (in meter squares)
Serum triglycerides | From enrollment to the end of treatment at 12 weeks
  Level of triglycerides fats in blood in measured in laboratory using venous blood sample
Total Cholesterol | From enrollment to the end of treatment at 12 weeks
  Level of total cholesterol in blood in measured in laboratory using venous blood sample
High Density Lipoproteins (HDL) | From enrollment to the end of treatment at 12 weeks
  High Density Lipoproteins (HDL) cholesterol fats are measured in laboratory using a venous blood sample
Low Density Lipoproteins (LDL) | From enrollment to the end of treatment at 12 weeks
  Low Density Lipoproteins (LDL) cholesterol fats are measured in laboratory using a venous blood sample

SECONDARY OUTCOMES:
HDL ratio | From enrollment to the end of treatment at 12 weeks
  The number of total cholesterol divided by high-density lipoprotein (HDL)

CONTACTS AND LOCATIONS:
Overall Officials: Radwa S Abdulrahman, PhD, Principal Investigator — Ass. Prof. Dept. of PT for Pediatric, Faculty of Physical Therapy, Badr University in Cairo, Egypt.; Hayam M Mahmoud, PhD, Study Chair — Professor Dept. of PT for Neurology & Neurosurgery, Faculty of Physical Therapy, Cairo Univ. Egypt; Wael OA Abd El-Khalek, PhD, Study Chair — Lecturer, Dept. of Basic Sciences, Faculty of Physical Therapy, Badr University in Cairo, Egypt.; Noha A Fouad, PhD, Study Chair — Ass Prof Dept. of PT for Women's Health Faculty of Physical Therapy Badr University in Cairo, Egyp; Mina AG Elias, PhD, Principal Investigator — Department of Physical Therapy Ahmed Maher Teaching hospital, General Organization For Teaching Hospitals And Institutes (GOTHI); Ashraf H Saleh, PhD, Study Chair — Prof Dept. of PT for Surgery and Burn, Faculty of Physical Therapy Badr University in Cairo, Egyp; Mona M Abdelkhalek, PhD, Study Chair — Ass. Prof. Dept. of PT for Internal Medicine, Faculty of Physical Therapy, Badr University in Cairo, Egypt.
Locations (2):
- Egypt (2):
  - Badr University in Cairo faculty of physical therapy, Cairo
  - El-Mahaba Specialized Charity Polyclinics., Cairo